CLINICAL TRIAL: NCT01944410
Title: Efficacy of Platelet-rich Plasma in Treatment of Mandibular Traumatic Bone Cyst
Brief Title: Use of PRP in Treatment of Mandibular Traumatic Bone Cyst
Acronym: TBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, oral and maxillofacial surgeon, Shiraz University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1234; 12345sums (Other Grant/Funding Number: shiraz university of medical sciences)
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Traumatic Bone Cyst
Keywords: PRP; TBC; Treatment
MeSH Terms: conditions — Bone Cysts | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- traumatic bone cyst (Experimental): Patients with traumatic bone cyst defect are injected with PRP
  Interventions: Biological: PRP injection

INTERVENTIONS:
Biological: PRP injection — injection of PRP to traumatic bone cyst defect
  Other Names: growth factor injection

SUMMARY:
The traumatic bone cyst (TBC) is an infrequent nonepithelial lined cavity of the jaws, which was first expressed by lucassin 1929, the lesion has attracted a great deal of interest in the dental literature, but its pathogenesis is still not evidently recognized. It determines a bone cavity of irregular shape which appears like a cyst on a radiograph, and histopathologically there are no elements to confirm a diagnosis of a cysts. TBC the international histological classification assumed by the World Health Organisation for odontogenic tumours utilizes the term "solitary bone cyst", nevertheless the term "traumatic bone cyst" (TBC) is more extensively used in the literature. The WHO classification explains TBC as a non-neoplastic osseous lesion because it demonstrates no epithelial lining, which differentiates this lesion from the true cysts. There is general conformity that most traumatic bone cysts present without symptoms or signs. Seldom, expansion of the cortical plate may occur with extraoral swelling, less commonly there may erosion through the cortical bone may take place.' Teeth in the area of involved bone usually remain vital, without root resorption or tooth mobility. Treatment of traumatic bone cysts has included surgical exploration and curettage to motivate bleeding within the bony cavity,' packing of the cyst cavity with Gelfoam which has been saturated with thrombin and penicillin, and bone grafting based on previous study Injection of autogeneic blood into the bony cavity of a traumatic bone cyst was followed by rapid resolution of the lesion.

Platelet-rich plasma (PRP) is a rich source of growth factors. The growth factors present in PRP are familiar, including transforming growth factor-_ (TGF-_1 and TGF-_2), vascular endothelial growth factor, 3 isomers of platelet-derived growth factor (PDGF-__,PDGF-__, and PDGF-__), and endothelial growth factor. These growth factors are considered to have the capacity to accelerate chemotaxis, mitogenesis, angiogenesis, and synthesis of collagen matrix and support tissue repair when applied on bone wounds. Due to this high platelet content, PRP has been used in orthopaedic surgery, oral implantology, and periodontics with the aim of making the repair process as fast and natural as possible, as it can potentially afford considerable tissue improvement in bone and soft tissue in a similar way. PRP is easily acquired, rich in cell signalling molecules, completely autogenous and can be obtained from minimal blood volumes.the purpose of the present study is to determine the efficacy of PRP in the treatment of mandibular TBC.

DETAILED DESCRIPTION:
The study sample consisted of 12 young adult volunteers presenting with TBC of mandible. Local ethical committee approval will be obtained before the trial starts. Laboratory tests (complete blood count, glucose, creatinine, platelets, lipid profile) were performed for all patients. These tests provided an important overview of patient health and a baseline for analysis of the prognosis of PRP use. The process for obtaining PRP basically consists of collection of a 20-mL sample of blood, centrifugation of this sample for 8 min, isolation of a 1-mL aliquot of plasma collected near the erythrocyte fraction. Surgical procedure includes: surgical exploration and injection of PRP to stimulate bone regeneration within the bony cavity . Bone repair was assessed by panoramic X-rays obtained at 2, 4, and 6 months postoperatively. Bone density was measured by area histogram analysis.

ELIGIBILITY:
Inclusion Criteria:

Traumatic Bone cyst diagnosed with panoramic X-Ray and histopathologic evaluation

* Intact cyst wall with high risk for fracture
* Patients of both sexes between 15 to 65 year's old
* Patients who are willing for evaluation in 2,4 and 6 months after surgery Patients who are willing for Laboratory tests . Provided written consent form
* Patients who agree to take xray in 2,4 and 6 months after surgery for radiographic evaluation

Exclusion Criteria:

* Patients who unable to undergo oral surgery
* Patients using systemic drugs or presenting a medical history positive for any systemic pathology history of hypersensitivity to any component used in the methodology Pregnant patients
* Smokers
* Patients who can not continue the study for private or social reasons

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Fulfill bone cyst defect | : 6 months
  change in size of the defect of bone will be measured by millimeter on radiographic examination in 2,4.6 months after PRP injection and will be compared with initial size of the defect

SECONDARY OUTCOMES:
effect of PRP | 6 months
  Evaluate effect of PRP injection to fulfill the defect of bone cyst and decrease size of the lesion

CONTACTS AND LOCATIONS:
Overall Officials: Reza Tabrizi, DMD, Study Chair — SUMS; Reza Tabrizi, DMD, Study Director — SUMS; Shole shahidi, DDS, Study Director — SUMS; Touba Karagah, DMD, Principal Investigator — SUMS; Nasibeh Zare, DDS, Principal Investigator — SUMS
Locations (1):
- RE, Shiraz, CMF Ward , Chamran Hospital , Chamran Avenue., Iran